CLINICAL TRIAL: NCT06986720
Title: Urdu Translation of Psychometric Properties Analysis of Revised High-Level Mobility Assessment Tool (HiMAT) in Healthy Children
Brief Title: Urdu Translation of Revised High-Level Mobility Assessment Tool (HiMAT) in Healthy Children
Status: Recruiting | Type: Observational
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Other Study IDs: REC/RCR&AHS/24/0729
Record Dates: First submitted 2025-05-15; First posted 2025-05-23 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Healthy Children
Keywords: revised HiMAT, Urdu translation, validation, mobility

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The ability to move with ease is labelled as mobility. Limitations in mobility are frequent, recovery of these skills is crucial for physical performance which gives children valuable social possibilities and has long-term advantages for their physical and mental health. The high-level mobility assessment tool (HiMAT) is a unidimensional performance to measure the degree of high-level mobility in traumatic brain injury patients. The revised HiMAT has been utilised recently in paediatric populations to assess clinical trial outcomes and measure high-level motor skills.

Urdu translation of revised HiMAT will be executed by using forward backwards translation method. Two bilingual translators fluent in both Urdu and English languages will facilitate the researcher in the translation of the tool. This final translated version will be then tested for validity and reliability on all participants of the study. The psychometric properties of the tool will be assessed including reliability, internal consistency, and item discrimination.

DETAILED DESCRIPTION:
Following steps will be followed for translation:

1. Forward Translation:

   Two independent translators who spoke Urdu as their native language will conduct initial translation into Urdu (U-HiMAT).
2. Synthesis:

   In this step both translated versions (U1 & U2) will be synthesized to obtain a common translated version of U-HiMAT. Full Urdu version of scale will be completed.
3. Backward Translation:

   Urdu translated version will be translated back into English by a different team consisting of professional independent bilingual translators.
4. Expert Committee:

   Expert committees consisting of pediatric physical therapists and pediatric clinical practitioners will evaluate and review the difference between a translated version and an original draft. They will create a pre final version for field testing.
5. Pre-Final Version Testing:

Pre-final Urdu and English version of scale will be tested on patients. Expert panel will review the findings from this process.

After completion of translation process, psychometric properties of the tool will be analysed.

ELIGIBILITY:
Inclusion Criteria:

* Children with age group 5-12 years
* No condition affecting mobility of children
* Able to understand and follow instruction.
* Can speak & understand language

Exclusion Criteria:

* Children with visual impairments.
* Children with conditions affecting their mobility.
* Children with any history of surgery in the past one year.
* Children with any cardiorespiratory comorbidities.
* Children with muscle strain, ligament sprain or joint laxity in lower extremities.
* Cognition less than 20 on Mini Mental State Examination (MMSE).
* Children with any history of any foot deformity

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The sample size is 80.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-05-12 (Actual); Primary Completion 2025-06-28 (Estimated); Study Completion 2025-07-16 (Estimated)

PRIMARY OUTCOMES:
Revised High Level Mobility Assessment Tool (HiMAT) | 6 months
  HiMAT is a single dimensional inspection of high-level movability for those suffering from TBI. The revised HiMAT comprises of 8 items that evaluate (1) walk forward, (2) walk backwards, (3) walk on toes and (4) walk over obstacle, (5) running, (6) skipping, (7) hopping, and (8) bounding. HiMAT has also been used to assess mobility in children with healthy conditions or suffering from any neurological disorder

CONTACTS AND LOCATIONS:
Overall Officials: Shazia Muheen, MS, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Williams G, Pallant J, Greenwood K. Further development of the High-level Mobility Assessment Tool (HiMAT). Brain Inj. 2010;24(7-8):1027-31. doi: 10.3109/02699052.2010.490517. PMID 20545456